CLINICAL TRIAL: NCT02130427
Title: A Volume, Motion, and Anatomically Adaptive Approach to Photon and Proton Beam Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC 08909
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Biopsy Proven Non Small Cell Lung Cancer; Head and Neck Cancer; Gastrointestinal Cancer; Colorectal Cancer; Rectal Cancers; Gynecological Malignancy Requiring Definitive Radiotherapy
Keywords: Adult subjects; NSCLC
MeSH Terms: conditions — Head and Neck Neoplasms; Gastrointestinal Neoplasms; Colorectal Neoplasms; Rectal Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lung Imaging (Other): Weekly 3D/4D CT scans during radiation therapy. MRI may be used in addition to or instead of CT depending on the location of the tumor and the decision of the treating physician.
  Interventions: Diagnostic Test: CT scan

INTERVENTIONS:
Diagnostic Test: CT scan — Weekly 3D/4D CT scan

SUMMARY:
This pilot study will determine changes over time in tumor volume/motion & patient anatomy, as well as dose distributions to normal organs. The study will inform medical decision-making about need for (and timing of) re-calibration of radiation dosimetry plans. Weekly CT and/or serial MR scans will be employed for those patients receiving 7-8 wks of radiation therapy. The study will enroll 30 patients in each stratum: Non small cell lung cancer (NSCLC), Head & Neck, gastrointestinal (GI) and Gynecologic tumor.

DETAILED DESCRIPTION:
This is a pilot study to estimate the degree of tumor volume, tumor motion and patient anatomy change during treatment with photon or proton beam radiotherapy. Patients will undergo simulation with an MR scan and/or CT scan per best clinical practices, and 4D imaging will be employed as indicated, at the discretion of the treating radiation oncologist. Photon beam treatment plans and Proton beam treatment plans will be generated from these images. Based on the location of the primary tumor, patients will undergo either up to weekly 3D or 4D CT and/or serial MR scans during treatment. These images will be compared to the initial CT/MR scans used for treatment planning and analyzed for changes in tumor volume and tumor anatomic location. At the end of treatment, the frequent 3D or 4D CT and/or serial MR images will be compared to the initial treatment planning images to quantify the changes in tumor volume and tumor motion during the course of radiation treatment. Each CT and/or MR Scan will also be used to evaluate the changes in dose distribution to the target volumes and normal tissues that occur with the initial photon treatment plan and initial proton treatment. The changes in tumor volume, tumor motion and dose distribution during the course of radiation treatment will be analyzed to determine the effect of tumor changes on radiation treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above.
* Biopsy proven diagnosis of non-small cell lung cancer, small cell lung cancer, head and neck, esophageal, gastric, pancreatic, anal, hepatic, biliary, colorectal, cervical, endometrial, vaginal, vulvar, ovarian cancer and any other gastrointestinal or gynecological cancers requiring definitive radiotherapy alone with or without concurrent chemotherapy.
* Able to provide written informed consent and comply with all study procedures.
* Entire course of radiotherapy will be delivered at the University of Pennsylvania Perelman Center for Advanced Medicine.

Exclusion Criteria:

- Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2022-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wei Zou, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Imaging: Weekly 3D/4D CT scans while receiving radiation therapy. Radiation therapy dosage metrics were not collected.
Period: Overall Study
Arm/Group | Imaging
Started | 74
Completed | 44
Not Completed | 30
Not completed — Imaging results not interpretable | 30

BASELINE CHARACTERISTICS:
Population: Only 44 Patients had interpretable GTV baseline measures from imaging
Groups:
- Imaging: Weekly 3D/4D CT scans; MRI scans used at the discretion of the treating physician when the location of the tumor requires it.
Arm/Group | Imaging
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Tumor volume [Mean (Standard Deviation); unit: cm^3] | 141.3 (158.4)

OUTCOME MEASURES:

1. Primary Outcome: Tumor Volume
Description: The degree of tumor volume, tumor motion and patient anatomy change during treatment with photon beam radiotherapy using 4D or 3D CT Scans and/or a serial of MR Imaging.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: cm^3
Groups:
- Completed Imaging: Weekly 3D/4D CT scans during radiation therapy. MRI may be used in addition to or instead of CT depending on the location of the tumor and the decision of the treating physician.
  CT scan: Weekly 3D/4D CT scan
Arm/Group | Completed Imaging
Number analyzed (Participants) | 44
cm^3 | 93.55 (63.77)

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this imaging trial.
Description: Adverse events were not collected for this imaging trial as they would not be relevant to the purposes of the trial (to track change in GTV over time via CT scans).
Groups:
- Complete Imaging: Weekly 3D/4D CT scans during radiation therapy. MRI may be used in addition to or instead of CT depending on the location of the tumor and the decision of the treating physician.
  CT scan: Weekly 3D/4D CT scan
Arm/Group | Complete Imaging
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT02130427/Prot_SAP_000.pdf